CLINICAL TRIAL: NCT03513458
Title: Late Phase Administration Anakinra as a Rescue Treatment for Inhaled Allergen Challenge-Induced Airway Inflammation
Acronym: LateAna
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: [The risk of inhaled allergen challenge and anakinra treatment outweigh benefits to participants with allergic asthma due to the COVID-19 pandemic.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 17-0779; 1R01HL135235-01A1 (NIH)
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Asthma
Keywords: Late Phase Asthmatic Response; Allergen Challenge
MeSH Terms: conditions — Asthma | interventions — Interleukin 1 Receptor Antagonist Protein; Receptors, Interleukin-6; Antigens, Dermatophagoides; Allergens

STUDY DESIGN:
Intervention Model Description: Subjects are randomized to one of two arms, either taking Anakinra or placebo. After a washout period, the subjects will be moved to the opposite arm.
Who Masked: Participant, Investigator
Masking Description: The randomization to study arms will be done by the department biostatistician and communicated to Investigational Drug Services to maintain the double-blind nature of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anakinra then Placebo (Experimental): Subjects randomized to this arm will receive the experimental treatment of Anakinra on their first exposure to Dermatophagoides Farinae (dust mite) allergen challenge, followed by the Anakinra matching placebo on their second exposure.
  Interventions: Biological: Anakinra; Other: Anakinra Matching Placebo; Drug: Dermatophagoides Farinae
- Placebo then Anakinra (Experimental): Subjects randomized to this arm will receive the inactive placebo on their first exposure to the Dust Mite Allergen challenge, followed by the experimental treatment of Anakinra on their second exposure.
  Interventions: Biological: Anakinra; Other: Anakinra Matching Placebo; Drug: Dermatophagoides Farinae

INTERVENTIONS:
Biological: Anakinra — A single 1mg/kg subcutaneous injection (up to 100 mg) of Anakinra will be administered at the onset of the LPR, roughly three hours post allergen challenge, to model Anakinra use in an emergency care setting.
  Other Names: Kinaret
Other: Anakinra Matching Placebo — A single dose of matching placebo will be administered at the onset of the LPR, roughly three hours post allergen challenge, to model Anakinra use in an emergency care setting.
  Other Names: dummy
Drug: Dermatophagoides Farinae — Standardized house dust mite Dermatophagoides farinae (D. farinae) allergen extract at 30,000 allergen units (AU)/mL for inhalation (provided by Greer Laboratories, Lenoir, NC).
  Other Names: Allergen extract

SUMMARY:
Purpose: The primary objective of this study is to examine the effectiveness of anakinra as a rescue treatment for allergic airway inflammation. Utilizing an inhaled allergen challenge model, the investigators will determine the effectiveness of a single 1 mg/kg dose of anakinra administered after inhaled allergen challenge for mitigating features of airway inflammation.

Participants: 25 mild allergic asthmatics sensitized to Dermatophagoides farinae (D. farinae) Procedures (methods): 12 eligible subjects of 25 volunteers will participate in a double blind cross-over study. Following randomization to the placebo or anakinra treatment group, subjects will undergo inhalation of D. farinae, and their early and late phase asthmatic responses will be measured. Subjects will undergo induced sputum sampling, methacholine challenge, and mucociliary clearance measures. After completion of period 1, subjects will cross over to the alternate study arm.

DETAILED DESCRIPTION:
Asthma is an increasingly common chronic illness with higher rates of hospitalization for exacerbation than many other chronic conditions. In 2009, total asthma costs in the U.S. were estimated at $56 billion per year, and over half the overall asthma-related costs were attributed to inpatient hospitalization. Allergen exposure and viral infection are among the most common triggers for asthma exacerbations. Exacerbations of allergic asthma are characterized by an early phase response (EPR), mediated by release of preformed mediators like histamine from mast cells, and a late phase response (LPR) 3-7 hours later mediated by chemokines and cytokines, including IL-1β, that attract leukocytes such as neutrophils and eosinophils to the airways, increase mucus production, trigger airway smooth muscle contraction, and result in airway constriction and airway hyper-reactivity (AHR). The LPR is thought to be predominantly responsible for the symptoms associated with acute exacerbations of allergic asthma.

While corticosteroids are considered a mainstay of treatment for asthma exacerbation regardless of the trigger, there are limitations to their effectiveness in the acute setting including the initial lag period of 4-6 hours or more before therapeutic effect and the concern for broad immune suppression. Corticosteroids are often ineffective in treating the neutrophilic component of airway inflammation seen with viral infection and allergen-induced airway inflammation . Finally, mucus plugging is a known hallmark of severe and fatal asthma, yet there is a notable lack of effective mucolytic treatments for asthma. Time to therapeutic benefit is key in preventing patient morbidity and mortality. Currently there is an urgent need for anti-inflammatory treatments that work quickly and effectively in acute asthma exacerbations.

The investigators propose that IL-1 blockade can achieve these ends and perhaps complement corticosteroid actions. Anakinra is an FDA-approved recombinant form of human IL-1 receptor antagonist (IL-1RA), a natural anti-inflammatory cytokine that competes with agonist binding to the IL-1 receptor, suppressing IL-1β and IL-1a signaling. Numerous studies indicate that IL-1 signaling mediates key features of viral- and allergen-induced airway inflammation. IL-1 signaling can directly impact three aspects of an airway inflammatory response: granulocyte (neutrophil/eosinophil) recruitment; non-specific and allergen-specific airway reactivity; and mucin production. Numerous IL-1 blocking agents are FDA-approved for conditions where the IL-1β pathway predominates disease pathophysiology, such as in systemic juvenile idiopathic arthritis and the cryopyrin-associated periodic syndromes.

Anakinra is an ideal candidate to test as a rescue treatment for acute asthma exacerbation due to its fast onset of action (reaching peak concentrations in 3-7 hours), and a short 4-6 hour half-life. A single 1mg/kg dose (up to 100mg) of anakinra or placebo will be administered at the onset of the LPR to model anakinra use in an emergency care setting. This dose was chosen because it is the current FDA-approved dose for rheumatoid arthritis (RA). Notably, the investigators have previously demonstrated that a 1 mg/kg dose resulted in significant reduction in airway granulocyte recruitment following lipopolysaccharide (LPS) challenge in a study of healthy volunteers. The investigators' objective is to determine if a single 1 mg/kg dose of Anakinra can mitigate key features of asthma exacerbations, namely AHR, airway constriction, airway inflammation, and mucous secretion/clearance.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-45 years, inclusive
* FEV1 of at least 80% of predicted and FEV1/FVC (forced vital capacity) ratio of at least 0.7 (without use of bronchodilator medications for 12 hours or long acting beta agonists for 24 hours), consistent with lung function of persons with no more than mild episodic or mild persistent asthma.
* Physician diagnosis of asthma
* Positive methacholine inhalation challenge as performed in the separate screening protocol within the prior 12 months (defined as provocative concentration of methacholine of 10 mg/mL or less producing a 20% fall in FEV1 (PC20 methacholine)
* Allergic sensitization to house dust mite (D. farinae) as confirmed by positive immediate skin prick test response
* Clinical reactivity to D. farinae assessed through inhaled allergen challenge with a decline in FEV1 of ≥20% from baseline in the early asthmatic response and ≥15% in the late asthmatic response.
* Negative pregnancy test for females who are not s/p hysterectomy with oophorectomy or who have not been amenorrheic for 12 months or more.
* Oxygen saturation of >94% and blood pressure within the following limits: (Systolic between 150-90 mmHg, Diastolic between 90-60 mmHg).
* Ability to provide an induced sputum sample.
* Negative intracutaneous tuberculin skin test (PPD) defined as less than 5mm induration for the purpose of this protocol (positive PPD contraindication to anakinra injection). A negative tuberculosis (TB) test within the past year (either PPD or quantiferon TB Gold) is also acceptable

Exclusion Criteria:

Clinical contraindications:

* Any chronic medical condition considered by the PI as a contraindication to participation in the study including significant cardiovascular disease, diabetes, chronic renal disease, chronic thyroid disease, history of chronic infections or immunodeficiency.
* Pregnancy or nursing a baby
* History of latex allergy/sensitivity
* Allergy/sensitivity to anakinra or its formulation
* Physician directed emergency treatment for an asthma exacerbation within the preceding 12 months.
* Exacerbation of asthma more than 2x/week which could be characteristics of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
* Daily requirements for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma (not to include prophylactic use of albuterol prior to exercise).
* Viral upper respiratory tract infection within 4 weeks of challenge.
* Any acute infection requiring antibiotics within 4 weeks of exposure or fever of unknown origin within 4 weeks of challenge.
* Severe asthma
* Mental illness of history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
* Cigarette smoking >1 pack per month
* Nighttime symptoms of cough or wheeze greater than 1x/week at baseline (not during a clearly recognized viral induced asthma exacerbation) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
* Allergy/sensitivity to study drugs or their formulations
* Known hypersensitivity to methacholine or to other parasympathomimetic agents
* History of intubation for asthma
* Unwillingness to limit coffee, tea, cola drinks, chocolate, or other foods containing caffeine after midnight on the days that methacholine challenge testing and inhaled allergen challenge is to be performed
* Unwillingness to use reliable contraception if sexually active (IUD, birth control pills/patch, condoms).
* Radiation history will be collected. Any subject whose exposure history within the past twelve months would cause them to exceed their annual limits will be excluded

Usage of the following medications:

* Use of systemic steroid therapy within the preceding 12 months for an asthma exacerbation. All use of systemic steroids in the last year will be reviewed by a study physician.
* Subjects who are prescribed daily inhaled corticosteroids, cromolyn, or leukotriene inhibitors (Montelukast or Zafirlukast) will be required to discontinue these medications at least 4 weeks prior to their screening visit.
* Use of daily theophylline within the past month.
* Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma. (Not to include prophylactic use of albuterol prior to exercise).
* Use of any immunosuppressant therapy within the preceding 12 months will be reviewed by the study physician.
* Use of any immunomodulatory therapy within the preceding 12 months.
* Use of beta blocking medications
* Antihistamines in the 5 days prior to allergen challenge
* Routine use of NSAIDs, including aspirin.

Physical/laboratory indications:

* Abnormalities on lung auscultation
* Temperature >37.8 C
* Oxygen saturation of <94%
* Systolic BP>150 mmHg or <90 mmHg or diastolic BP>90 mmHg or <60 mmHg
* Absolute neutrophil count <1.4 x 109/L

Inability or unwillingness of a participant to give written informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Maximum % FEV1 drop from Baseline during LPR period | Baseline and 3-10 hours following PD20
  The principal endpoint will be maximal % drop in Forced Expiratory Volume in 1 second (FEV1) from baseline during the LPR period (3-10 hours). The FEV1 following saline and prior to the first dose of antigen during the inhaled allergen challenge will be considered the baseline value. Declines in FEV1 will be measured as a % drop from the baseline. A provocative dose causing a 20% fall FEV1 (PD20) is determined during the allergen challenge.

SECONDARY OUTCOMES:
Area under the curve (AUC) measuring % drop in FEV1 in the LPR | Baseline and 3-10 hours following PD20
  The FEV1 following saline and prior to the first dose of antigen during the inhaled allergen challenge will be considered the baseline value from which the % drop in FEV1 will be determined.
Change in Methacholine reactivity, as measured by the concentration of methacholine resulting in a 20% drop in FEV1 (PC20) | Baseline and 24 hours post allergen challenge
  Participants will undergo a methacholine challenge to assess airway hyper-responsiveness at baseline. Change in methacholine reactivity, as measured by the PC20, from baseline to 24 hours after the allergen challenge will be determined.
Fractional exhaled Nitric Oxide (FeNO) as an exploratory biomarker | Baseline and 24 hours post allergen challenge
  FeNO is being investigated as a non-invasive airway inflammation marker. FeNO is measured in ppb with a chemoluminescence analyzer before the saline and prior to the first dose of antigen during the inhaled allergen challenge and at 24 hours post the allergen challenge.
Change in % eosinophils in induced sputum | Baseline and 24 hours post allergen challenge
  An induced sputum sample will be processed and counted to provide the % change in eosinophils between the two time points.
Change in % neutrophils in induced sputum | Baseline and 24 hours post allergen challenge
  An induced sputum sample will be processed and counted to provide the % change in neutrophils between the two time points.
Change in eosinophils per mg of induced sputum | Baseline and 24 hours post allergen challenge
  An induced sputum sample will be processed and counted to provide the eosinophils per mg change between the two time points.
Change in neutrophils per mg of induced sputum | Baseline and 24 hours post allergen challenge
  An induced sputum sample will be processed and counted to provide the neutrophils per mg change between the two time points.
Change in Sputum levels of major respiratory mucin MUC5AC | Baseline and 24 hours post allergen challenge
  An induced sputum sample will be processed and analyzed for the amount of protein MUC5AC between the two time points.
Change in Sputum levels of major respiratory mucin MUC5B | Baseline and 24 hours post allergen challenge
  An induced sputum sample will be processed and analyzed for the amount of protein MUC5B between the two time points.
Change in Mucociliary clearance (MCC) | 4 hours post allergen challenge
  The change in MCC will be measured as % tracheobronchial retention of radiolabeled particles in the airways.
Central (C) vs. peripheral (P) deposition ratio (C/P) | 4 hours post allergen challenge
  C/P is a reflection of deposition in the central airways during MCC.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hernandez, MD, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: No
The investigators will not be sharing individual participant data (IPD) with other researchers.

REFERENCES:
- [Background] Moorman JE, Akinbami LJ, Bailey CM, Zahran HS, King ME, Johnson CA, Liu X. National surveillance of asthma: United States, 2001-2010. Vital Health Stat 3. 2012 Nov;(35):1-58. PMID 24252609
- [Background] Kaur BP, Lahewala S, Arora S, Agnihotri K, Panaich SS, Secord E, Levine D. Asthma: Hospitalization Trends and Predictors of In-Hospital Mortality and Hospitalization Costs in the USA (2001-2010). Int Arch Allergy Immunol. 2015;168(2):71-8. doi: 10.1159/000441687. Epub 2015 Nov 24. PMID 26595589
- [Background] Bahadori K, Doyle-Waters MM, Marra C, Lynd L, Alasaly K, Swiston J, FitzGerald JM. Economic burden of asthma: a systematic review. BMC Pulm Med. 2009 May 19;9:24. doi: 10.1186/1471-2466-9-24. PMID 19454036
- [Background] Hasegawa K, Tsugawa Y, Brown DF, Camargo CA Jr. Childhood asthma hospitalizations in the United States, 2000-2009. J Pediatr. 2013 Oct;163(4):1127-33.e3. doi: 10.1016/j.jpeds.2013.05.002. Epub 2013 Jun 12. PMID 23769497
- [Background] Jackson DJ, Sykes A, Mallia P, Johnston SL. Asthma exacerbations: origin, effect, and prevention. J Allergy Clin Immunol. 2011 Dec;128(6):1165-74. doi: 10.1016/j.jaci.2011.10.024. PMID 22133317
- [Background] Stoppelenburg AJ, Salimi V, Hennus M, Plantinga M, Huis in 't Veld R, Walk J, Meerding J, Coenjaerts F, Bont L, Boes M. Local IL-17A potentiates early neutrophil recruitment to the respiratory tract during severe RSV infection. PLoS One. 2013 Oct 23;8(10):e78461. doi: 10.1371/journal.pone.0078461. eCollection 2013. PMID 24194936
- [Background] Zhu J, Message SD, Qiu Y, Mallia P, Kebadze T, Contoli M, Ward CK, Barnathan ES, Mascelli MA, Kon OM, Papi A, Stanciu LA, Jeffery PK, Johnston SL. Airway inflammation and illness severity in response to experimental rhinovirus infection in asthma. Chest. 2014 Jun;145(6):1219-1229. doi: 10.1378/chest.13-1567. PMID 24457412
- [Background] Grunberg K, Smits HH, Timmers MC, de Klerk EP, Dolhain RJ, Dick EC, Hiemstra PS, Sterk PJ. Experimental rhinovirus 16 infection. Effects on cell differentials and soluble markers in sputum in asthmatic subjects. Am J Respir Crit Care Med. 1997 Aug;156(2 Pt 1):609-16. doi: 10.1164/ajrccm.156.2.9610079. PMID 9279247
- [Background] Nagarkar DR, Bowman ER, Schneider D, Wang Q, Shim J, Zhao Y, Linn MJ, McHenry CL, Gosangi B, Bentley JK, Tsai WC, Sajjan US, Lukacs NW, Hershenson MB. Rhinovirus infection of allergen-sensitized and -challenged mice induces eotaxin release from functionally polarized macrophages. J Immunol. 2010 Aug 15;185(4):2525-35. doi: 10.4049/jimmunol.1000286. Epub 2010 Jul 19. PMID 20644177
- [Background] Fanta CH, Rossing TH, McFadden ER Jr. Glucocorticoids in acute asthma. A critical controlled trial. Am J Med. 1983 May;74(5):845-51. doi: 10.1016/0002-9343(83)91076-8. PMID 6340496
- [Background] Ellul-Micallef R. The acute effects of corticosteroids in bronchial asthma. Eur J Respir Dis Suppl. 1982;122:118-25. PMID 6958475
- [Background] Scarfone RJ, Fuchs SM, Nager AL, Shane SA. Controlled trial of oral prednisone in the emergency department treatment of children with acute asthma. Pediatrics. 1993 Oct;92(4):513-8. PMID 8414819
- [Background] Stuck AE, Minder CE, Frey FJ. Risk of infectious complications in patients taking glucocorticosteroids. Rev Infect Dis. 1989 Nov-Dec;11(6):954-63. doi: 10.1093/clinids/11.6.954. PMID 2690289
- [Background] Ulich TR, Yin SM, Guo KZ, del Castillo J, Eisenberg SP, Thompson RC. The intratracheal administration of endotoxin and cytokines. III. The interleukin-1 (IL-1) receptor antagonist inhibits endotoxin- and IL-1-induced acute inflammation. Am J Pathol. 1991 Mar;138(3):521-4. PMID 1825745
- [Background] Hudock KM, Liu Y, Mei J, Marino RC, Hale JE, Dai N, Worthen GS. Delayed resolution of lung inflammation in Il-1rn-/- mice reflects elevated IL-17A/granulocyte colony-stimulating factor expression. Am J Respir Cell Mol Biol. 2012 Oct;47(4):436-44. doi: 10.1165/rcmb.2012-0104OC. Epub 2012 May 16. PMID 22592923
- [Background] Tsukagoshi H, Sakamoto T, Xu W, Barnes PJ, Chung KF. Effect of interleukin-1 beta on airway hyperresponsiveness and inflammation in sensitized and nonsensitized Brown-Norway rats. J Allergy Clin Immunol. 1994 Feb;93(2):464-9. doi: 10.1016/0091-6749(94)90355-7. PMID 8120273
- [Background] Barchasz E, Naline E, Molimard M, Moreau J, Georges O, Emonds-Alt X, Advenier C. Interleukin-1beta-induced hyperresponsiveness to [Sar9,Met(O2)11]substance P in isolated human bronchi. Eur J Pharmacol. 1999 Aug 20;379(1):87-95. doi: 10.1016/s0014-2999(99)00484-7. PMID 10499376
- [Background] Wang CC, Fu CL, Yang YH, Lo YC, Wang LC, Chuang YH, Chang DM, Chiang BL. Adenovirus expressing interleukin-1 receptor antagonist alleviates allergic airway inflammation in a murine model of asthma. Gene Ther. 2006 Oct;13(19):1414-21. doi: 10.1038/sj.gt.3302798. Epub 2006 May 25. PMID 16724092
- [Background] Okada S, Inoue H, Yamauchi K, Iijima H, Ohkawara Y, Takishima T, Shirato K. Potential role of interleukin-1 in allergen-induced late asthmatic reactions in guinea pigs: suppressive effect of interleukin-1 receptor antagonist on late asthmatic reaction. J Allergy Clin Immunol. 1995 Jun;95(6):1236-45. doi: 10.1016/s0091-6749(95)70081-1. PMID 7797792
- [Background] Chen Y, Garvin LM, Nickola TJ, Watson AM, Colberg-Poley AM, Rose MC. IL-1beta induction of MUC5AC gene expression is mediated by CREB and NF-kappaB and repressed by dexamethasone. Am J Physiol Lung Cell Mol Physiol. 2014 Apr 15;306(8):L797-807. doi: 10.1152/ajplung.00347.2013. Epub 2014 Jan 31. PMID 24487386
- [Background] Evans CM, Raclawska DS, Ttofali F, Liptzin DR, Fletcher AA, Harper DN, McGing MA, McElwee MM, Williams OW, Sanchez E, Roy MG, Kindrachuk KN, Wynn TA, Eltzschig HK, Blackburn MR, Tuvim MJ, Janssen WJ, Schwartz DA, Dickey BF. The polymeric mucin Muc5ac is required for allergic airway hyperreactivity. Nat Commun. 2015 Feb 17;6:6281. doi: 10.1038/ncomms7281. PMID 25687754
- [Background] Garlanda C, Dinarello CA, Mantovani A. The interleukin-1 family: back to the future. Immunity. 2013 Dec 12;39(6):1003-18. doi: 10.1016/j.immuni.2013.11.010. PMID 24332029
- [Background] Hernandez ML, Mills K, Almond M, Todoric K, Aleman MM, Zhang H, Zhou H, Peden DB. IL-1 receptor antagonist reduces endotoxin-induced airway inflammation in healthy volunteers. J Allergy Clin Immunol. 2015 Feb;135(2):379-85. doi: 10.1016/j.jaci.2014.07.039. Epub 2014 Sep 5. PMID 25195169